CLINICAL TRIAL: NCT04263844
Title: Comparison of Efficacy of Premedication Between Dexmedetomidine and Midazolam Intranasal for the Prevention of Emergence Delirium in Children Undergoing Ophthalmic Surgery
Brief Title: Intranasal Dexmedetomidine Versus Intranasal Midazolam for Emergence Delirium Prevention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Andi Ade Wijaya Ramlan, Principal Investigator, Pediatric Anesthesia Division, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IndonesiaUAnes 051
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Emergence Delirium
Keywords: emergence, delirium, dexmedetomidine, midazolam, pediatric
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Active Comparator): subject will receive premedication with intranasal dexmedetomidine 1 mcg/kgBB thirty minutes before induction
  Interventions: Drug: Intranasal dexmedetomidine
- Midazolam (Active Comparator): subject will receive premedication with intranasal midazolam 0,1 mg/kgBB thirty minutes before induction
  Interventions: Drug: Intranasal Midazolam

INTERVENTIONS:
Drug: Intranasal dexmedetomidine — subject will receive premedication with intranasal dexmedetomidine thirty minutes before induction
  Arms: Dexmedetomidine
Drug: Intranasal Midazolam — subject will receive premedication with intranasal midazolam thirty minutes before induction
  Arms: Midazolam

SUMMARY:
This study is a double-blind clinical trial, in pediatric patients aged 1-12 years with physical status ASA (American Society of Anesthesiology) 1 and 2 who underwent eye surgery under general anesthesia using Sevoflurane inhalation agents, in investigator institution during February-May 2019.. There were 64 children obtained by consecutive sampling, who underwent eye surgery in investigator institution during February-May 2019. The subjects then grouped into dexmedetomidine group and midazolam group. Effectiveness was assessed from Emergence Delirium (ED) events, recovery time, and post-premedication desaturation events. Data analysis using Chi Square test and Mann-Whitney test.

DETAILED DESCRIPTION:
There were 64 children obtained by consecutive sampling, The subjects then grouped into dexmedetomidine group and midazolam group. Effectiveness was assessed from ED events, recovery time, and post-premedication desaturation events.

ELIGIBILITY:
Inclusion Criteria:

* children undergoing ophthalmologic surgery with general anesthesia
* children aged 1 - 12 years old
* physical status ASA 1-2
* signing informed consent

Exclusion Criteria:

* children undergoing emergency surgery
* children with PICU nursing after surgery
* children with psychological and neurological condition
* children with allergic history to dexmedetomidine and midazolam
* children with history of malignant hyperthermia or family history of malignant hyperthermia
* children with possibility of difficult intubation and ventilation

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
incidence of emergence delirium thirty minutes after surgery | 30 minutes
  PAED score was measured

CONTACTS AND LOCATIONS:
Overall Officials: Andi Ade W Ramlan, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cohen MM, Cameron CB, Duncan PG. Pediatric anesthesia morbidity and mortality in the perioperative period. Anesth Analg. 1990 Feb;70(2):160-7. doi: 10.1213/00000539-199002000-00005. PMID 2301747
- [Result] Mohkamkar M Bs, Farhoudi F Md, Alam-Sahebpour A Md, Mousavi SA Md, Khani S PhD, Shahmohammadi S BSc. Postanesthetic Emergence Agitation in Pediatric Patients under General Anesthesia. Iran J Pediatr. 2014 Apr;24(2):184-90. PMID 25535538
- [Result] Kim JH. Mechanism of emergence agitation induced by sevoflurane anesthesia. Korean J Anesthesiol. 2011 Feb;60(2):73-4. doi: 10.4097/kjae.2011.60.2.73. Epub 2011 Feb 25. No abstract available. PMID 21390159
- [Result] Silva LM, Braz LG, Modolo NS. Emergence agitation in pediatric anesthesia: current features. J Pediatr (Rio J). 2008 Mar-Apr;84(2):107-13. doi: 10.2223/JPED.1763. PMID 18372935
- [Result] Key KL, Rich C, DeCristofaro C, Collins S. Use of propofol and emergence agitation in children: a literature review. AANA J. 2010 Dec;78(6):468-73. PMID 21309294
- [Result] Lee CJ, Lee SE, Oh MK, Shin CM, Kim YJ, Choe YK, Cheong SH, Lee KM, Lee JH, Lim SH, Kim YH, Cho KR. The effect of propofol on emergence agitation in children receiving sevoflurane for adenotonsillectomy. Korean J Anesthesiol. 2010 Aug;59(2):75-81. doi: 10.4097/kjae.2010.59.2.75. Epub 2010 Aug 20. PMID 20740210